CLINICAL TRIAL: NCT02016365
Title: A Phase II Multicenter Pilot Study of the Safety and Efficacy of Doxycycline/UrsoDeoxyCholicAcid on Disease Progression in ATTR Amyloidosis
Brief Title: Safety and Efficacy Study of Doxycycline/UrsoDeoxyCholicAcid on Disease Progression in ATTR Amyloidosis
Acronym: Dox/Urso
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Ole B Suhr, Professor, MD, PhD, Professor, MD, PhD, Umeå University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT No:2011-005236-25
Record Dates: First submitted 2012-04-19; First posted 2013-12-20 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Transthyretin Amyloidosis; Cardiomyopathy
Keywords: Transthyretin amyloidosis; Cardiomyopathy; ATTR; neuropathy
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Cardiomyopathies | interventions — Doxycycline; Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doxycycline and UDCA (Experimental): Doxycycline (200 mg/day intermittently) and UDCA (750 mg/day continuously)
  Interventions: Drug: Doxycycline; Drug: Ursodeoxycholic acid

INTERVENTIONS:
Drug: Doxycycline — 200 mg/day (100 mg twice daily, orally) for 4 weeks with a pause of 2 weeks in combination with UDCA
  Other Names: Doxyferm
Drug: Ursodeoxycholic acid — 750 mg/day (500 mg +250mg orally) continuously
  Other Names: Ursofalk

SUMMARY:
The primary objective for this study is to evaluate the efficacy of doxycycline + ursodeoxycholic acid (UDCA) on disease progression in Transthyretin Amyloidosis (ATTR) subjects with cardiomyopathy with or without neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Cardiomyopathy with septal thickness > 15 mm and/or S-NT-ProBNP > 300 ng/
* Age >50 years
* Male and females after menopause. Menopause is defined as 6 to 12 months of amenorrhea in a woman over 45 years of age.
* Written informed consent to be obtained prior to any study procedure
* Histochemical diagnosis of amyloidosis as based on detection by polarizing microscopy of green birefringent material in Congo red-stained tissue specimens, and typing of amyloid deposits as TTR and identification of amyloid fibril type.
* Molecular definition of the TTR mutation or immunohistochemical staining of amyloid fibrils with anti TTR antibody
* New York Heart Association (NYHA) class <III
* Systolic blood pressure >100 mmHg (standing)
* Must have symptomatic organ involvement with amyloid to justify therapy

Exclusion Criteria:

* Liver transplantation in the previous 6 months or liver transplantation anticipated in less than 6 months;
* ALT and/or AST > 2 x upper normal limit (UNL);
* Creatinine clearance < 30 ml/min (Cockcroft -Gault Formula)
* Any other lab values, illness or condition that in the opinion of the investigator might place the subject at unacceptable risk for participation in the study;
* History of hypersensitivity to any of the ingredients of the study therapies;
* Use of any investigational drug, device (or biologic) within 4 weeks prior to study entry or during the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The efficacy on serum N terminal proBNP (NT-proBNP) | At 12 month treatment
  The primary endpoint of the study is the response rate to doxycycline + UDCA treatment at month 12. A responder is an ATTR subject with:
  - a reduction of, or an increase in serum NT-proBNP concentration of less than 30% of pre-treatment level will be regarded as consistent with treatment efficacy

SECONDARY OUTCOMES:
Modified Body Mass Index (mBMI) reduction | 12 month
  mBMI-reduction of less than 10%
Increase of septum thickness | 12 month
  Increase of septum thickness ≤ 2 mm
Neurologic Kumamoto Scale | 6, 12 and 18 month
  To assess the change from baseline in the neurologic Kumamoto Scale
Number of patients with adverse events | During 12 month treatment and during 6 month follow-up
  To assess the tolerability and safety of the treatment, the number of patients with adverse reactions will be recorded.
  Monthly phone contacts will be performed for monitoring of the treatment safety.
  The safety profile of doxycycline + UDCA will be assessed through the recording, reporting and analysis of baseline medical conditions, physical examination findings including vital signs and laboratory tests. These will be compared to analysis results observed during the study.
Blood work for potential drug-related adverse events | 18 months
  To assess the tolerability and safety of the treatment, blood work [e.g.complete blood count, creatinine and aspartate transaminase (AST), alkaline phosphatase(ALT)] for potential drug-related adverse events will be drawn at 1, 3, 6, 9, 12 and 18 month.
  The safety profile of doxycycline + UDCA will be assessed through the recording, reporting and analysis of baseline medical conditions, physical examination findings including vital signs and laboratory tests. These will be compared to analysis results observed during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ole B Suhr, MD PhD Prof, Principal Investigator — Dept of Clinical Medicine and public Health, Umeå University
Locations (3):
- Sweden (3):
  - Dept of Clinical Medicin, Ptieå Hospital, Piteå
  - Dept of clinical medicin, Skellefteå Hospital, Skellefteå
  - Dept of Clinical Medicine, Umeå University Hospital, Umeå